CLINICAL TRIAL: NCT04305288
Title: Modified FOLFIRINOX Versus Gemcitabine Plus Oxaliplatin as First-line Chemotherapy for Patients With Locally Advanced or Metastatic Cholangiocarcinoma
Brief Title: Chemotherapy mFOLFIRINOX in Locally Advanced or Metastatic Cholangiocarcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Yingbin Liu, MD, PhD, FACS, head of general surgery department，xin hua Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: CCA20191021
Record Dates: First submitted 2020-03-10; First posted 2020-03-12 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Cholangiocarcinoma of the Bile Duct

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gemox: The patients received conventional chemotherapy Gemox
- mFOLFIRINOX: The patients received chemotherapy modified FOLFIRINOX

SUMMARY:
The aim of this study was to evaluate the effectiveness of modified FOLFIRINOX (mFOLFIRINOX) compared to that of gemcitabine plus oxaliplatin (Gemox) for patients with locally advanced or metastatic CCA

DETAILED DESCRIPTION:
The aim of this study was to evaluate the effectiveness of modified FOLFIRINOX (mFOLFIRINOX) compared to that of gemcitabine plus oxaliplatin (Gemox) for patients with locally advanced or metastatic CCA

ELIGIBILITY:
The inclusion criteria included: patients aged 18-70 years old, regardless of gender; patients with locally advanced or metastatic CCA diagnosed by imaging and pathology; modified FOLFIRINOX regimen or Gemox regimen as first-line treatment; ≥ 1 focus that can be evaluated by imaging examination.

Exclusion criteria included: incomplete clinical history data; suffering from other malignant tumors within 5 years, except basal cell carcinoma and cervical carcinoma in situ; having received other systemic chemotherapy, targeted therapy, immunotherapy or radiotherapy as first-line treatment; with severe organ dysfunction.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced or metastatic CCA.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | up to 1 year
  From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 year. The progression is defined consistent with Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria for solid tumors.

SECONDARY OUTCOMES:
Overall survival | up to 2 years
Objective Response Rate | up to 1 year
  Objective Response Rate is defined as the percentage of patients with a complete or partial response to treatment,consistent with RECIST version 1.1 criteria for solid tumors.
Disease Control Rate | up to 1 year
  Disease Control Rate is defined as the percentage of patients with a complete or partial response to treatment or stable disease, consistent with RECIST version 1.1 criteria for solid tumors.
percentage of patients with Clinical Benefit Response | up to 1 year
  Composite measure based on patient-reported pain (per Faces pain scale revised), patient-reported pain medication, Karnofsky performance status(KPS), and weight. Clinical benefit is indicated by either:(a) improvement in pain (less pain intensity with stable or decreased pain medication; or less pain medication with stable or decreased pain intensity with stable or improved KPS; or (b) improvement in KPS with stable or improved pain.With stable for KPS and pain, clinical benefit may be indicated with an observation of positive weight change.
  Clinical benefit response (CBR) was classified weekly and a patient was considered a clinical benefit responder if clinical benefit was observed and maintained over a 4 week period.

CONTACTS AND LOCATIONS:
Overall Officials: yingbin liu, PHD, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xinhua Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zou L, Li X, Wu X, Cui J, Cui X, Song X, Ren T, Han X, Zhu Y, Li H, Wu W, Wang X, Gong W, Wang L, Li M, Lau WY, Liu Y. Modified FOLFIRINOX versus gemcitabine plus oxaliplatin as first-line chemotherapy for patients with locally advanced or metastatic cholangiocarcinoma: a retrospective comparative study. BMC Cancer. 2021 Jul 16;21(1):818. doi: 10.1186/s12885-021-08549-2. PMID 34266407